CLINICAL TRIAL: NCT01808573
Title: A STUDY OF NERATINIB PLUS CAPECITABINE VERSUS LAPATINIB PLUS CAPECITABINE IN PATIENTS WITH HER2+ METASTATIC BREAST CANCER WHO HAVE RECEIVED TWO OR MORE PRIOR HER2-DIRECTED REGIMENS IN THE METASTATIC SETTING (NALA)
Brief Title: A Study of Neratinib Plus Capecitabine Versus Lapatinib Plus Capecitabine in Patients With HER2+ Metastatic Breast Cancer Who Have Received Two or More Prior HER2 Directed Regimens in the Metastatic Setting
Acronym: NALA
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Puma Biotechnology, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PUMA-NER-1301; 2012-004492-38 (EudraCT Number); UTN U1111-1161-1603 (Other: WHO)
Record Dates: First submitted 2013-03-04; First posted 2013-03-11 (Estimated); Results first posted 2019-12-11 (Actual); Last update posted 2021-06-11 (Actual); Status verified 2021-05

CONDITIONS: HER2+ Metastatic Breast Cancer (MBC)
Keywords: Neratinib; Nerlynx
MeSH Terms: interventions — neratinib; Capecitabine; Lapatinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- neratinib plus capecitabine (Experimental): neratinib 240 mg orally, once daily with food, continuously in 21 day cycles, and capecitabine 1500 mg/m^2 daily in 2 evenly divided doses, orally with water within 30 minutes after a meal, taken on days 1 to 14 of each 21 day cycle.
  Interventions: Drug: neratinib; Drug: capecitabine
- lapatinib plus capecitabine (Active Comparator): lapatinib 1250 mg orally, once daily, continuously in 21 day cycles, and capecitabine 2000 mg/m^2 daily in 2 evenly divided doses, orally with water within 30 minutes after a meal, taken on days 1 to 14 of each 21 day cycle.
  Interventions: Drug: capecitabine; Drug: lapatinib

INTERVENTIONS:
Drug: neratinib
  Other Names: Nerlynx
  Arms: neratinib plus capecitabine
Drug: capecitabine
  Other Names: Xeloda
Drug: lapatinib
  Other Names: Tykerb; Tyverb
  Arms: lapatinib plus capecitabine

SUMMARY:
This is a randomized, multi-center, multinational, open-label, active-controlled, parallel design study of the combination of neratinib plus capecitabine versus the combination of lapatinib plus capecitabine in HER2+ MBC patients who have received two or more prior HER2 directed regimens in the metastatic setting.

DETAILED DESCRIPTION:
This is a randomized, multi-center, multinational, open-label, active-controlled, parallel design study of the combination of neratinib plus capecitabine versus the combination of lapatinib plus capecitabine in HER2+ MBC patients who have received two or more prior HER2 directed regimens in the metastatic setting. Patients will be randomized in a 1:1 ratio to one of the following treatment arms:

* Arm A: neratinib (240 mg once daily) + capecitabine (1500 mg/m^2 daily, 750 mg/m^2 twice daily [BID])
* Arm B: lapatinib (1250 mg once daily) + capecitabine (2000 mg/m^2 daily, 1000 mg/m^2 BID)

Patients will receive either neratinib plus capecitabine combination or lapatinib plus capecitabine combination until the occurrence of death, disease progression, unacceptable toxicity, or other specified withdrawal criterion.

ELIGIBILITY:
Inclusion Criteria:

* Aged ≥18 years at signing of informed consent.
* Histologically confirmed MBC, current stage IV.
* Documented HER2 overexpression or gene-amplified tumor immunohistochemistry 3+ or 2+, with confirmatory fluorescence in situ hybridization (FISH) +.
* Prior treatment with at least two (2) HER2-directed regimens for metastatic breast cancer.

Exclusion Criteria:

* Received previous therapy with capecitabine, neratinib, lapatinib, or any other HER2 directed tyrosine kinase inhibitor.

Note: There are additional inclusion and exclusion criteria. The study center will determine if you meet all of the criteria.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 621 (Actual)
Dates: Start 2013-03-29 (Actual); Primary Completion 2018-09-28 (Actual); Study Completion 2019-12-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Senior Vice President Clinical Science and Pharmacology, Study Director — Puma Biotechnology, Inc.
Locations (250):
- United States (77):
  - Ironwood Cancer and Research Centers, Chandler, Arizona
  - Ironwood Cancer and Research Centers, Gilbert, Arizona
  - Ironwood Cancer and Research Centers, Mesa, Arizona
  - Ironwood Cancer and Research Centers, Scottsdale, Arizona
  - UCLA Hematology Oncology, Alhambra, California
  - CBCC Global Research, Inc. at Comprehensive Blood and Caner Center, Bakersfield, California
  - Compassionate Cancer Care Medical Group Inc., Fountain Valley, California
  - St. Jude Heritage Medical Group, Fullerton, California
  - Marin Cancer Care, Inc., Greenbrae, California
  - UCLA Hematology Oncology, Irvine, California
  - University of California San Diego Medical Center, La Jolla, California
  - University of California San Diego Moores Cancer Center, La Jolla, California
  - Breastlink Medical Group, Inc., Orange, California
  - UCLA Hematology Oncology, Pasadena, California
  - UCLA Hematology Oncology, Porter Ranch, California
  - Emad Ibrahim, MD, Redlands, California
  - Cancer Care Associates Medical Group, Inc, Redondo Beach, California
  - Compassionate Cancer Care Medical Group, Riverside, California
  - University of California San Diego Medical Center - Hillcrest, San Diego, California
  - Sharp Memorial Hospital, San Diego, California
  - Breastlink Medical Group, Inc., Santa Ana, California
  - Cancer Center of Santa Barbara Sansum Clinic, Santa Barbara, California
  - Central Coast Medical Oncology, Santa Maria, California
  - UCLA Hematology Oncology, Santa Monica, California
  - Cancer Center of Santa Barbara, Solvang, California
  - UCLA Healthcare Santa Clarita Oncology, Valencia, California
  - UCLA Hematology/Oncology, Westlake Village, California
  - Sibley Memorial Hospital, Washington D.C., District of Columbia
  - Broward Medical Oncology Office, Plantation, Florida
  - Florida Cancer Research Institute, Plantation, Florida
  - Emory University Hospital Midtown, Atlanta, Georgia
  - Emory Clinic, Atlanta, Georgia
  - Emory University Winship Cancer Institute, Atlanta, Georgia
  - OnCare Hawaii, Honolulu, Hawaii
  - Queen's Medical Center, Honolulu, Hawaii
  - Straub Clinic and Hospital, Honolulu, Hawaii
  - University of Hawaii Cancer Center, Honolulu, Hawaii
  - Resurrection Medical Group, Chicago, Illinois
  - North Shore Oncology-Hematology Associates, Ltd., Crystal Lake, Illinois
  - Primary Healthcare Associates, SC, Harvey, Illinois
  - North Shore Hematology Oncology, Highland Park, Illinois
  - North Shore Oncology-Hematology Associates, Ltd., Libertyville, Illinois
  - Orchard Healthcare Research Inc, Skokie, Illinois
  - Primary Health Oncology, Hobart, Indiana
  - St. Mary Medical Center, Hobart, Indiana
  - Community Hospital, Munster, Indiana
  - Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins Hospital, Baltimore, Maryland
  - Sidney Kimmel Comprehensive Cancer Center at John Hopkins at Greenspring Station, Lutherville, Maryland
  - The Cancer Institute at University of Maryland St. Joseph Medical Center, Towson, Maryland
  - Massachusetts General Hospital, Boston, Massachusetts
  - Dana Farber Cancer Institute, Boston, Massachusetts
  - Karmanos Cancer Institute, Detroit, Michigan
  - Siteman Cancer Center - St. Peters, City of Saint Peters, Missouri
  - Washington University in St. Louis, St Louis, Missouri
  - Siteman Cancer Center - South County, St Louis, Missouri
  - Siteman Cancer Center - West County, St Louis, Missouri
  - Cancer Institute of New Jersey, New Brunswick, New Jersey
  - North Shore Hematology Oncology Association PC, East Setauket, New York
  - Clinical Research Alliance, Lake Success, New York
  - NYU Langone Medical Center, Lake Success, New York
  - Clinical Research Alliance, Inc., New York, New York
  - Weill Cornell Medical College, New York, New York
  - University Hospitals Cleveland Medical Center, Cleveland, Ohio
  - Cleveland Clinic Taussig Cancer Center, Cleveland, Ohio
  - University Hospitals Case Medical Center, Orange, Ohio
  - UPMC Cancer Pavillion, Greensburg, Pennsylvania
  - Hershey Medical Center, Hershey, Pennsylvania
  - UPMC Cancer Pavillion, Monroeville, Pennsylvania
  - Magee Women's Hospital, Pittsburgh, Pennsylvania
  - UPMC Cancer Pavillion, Pittsburgh, Pennsylvania
  - Hillman Cancer Center, Pittsburgh, Pennsylvania
  - UPMC Cancer Pavillion, Uniontown, Pennsylvania
  - UPMC Cancer Pavillion, West Mifflin, Pennsylvania
  - West Clinic PC, Germantown, Tennessee
  - West Clinic PC, Memphis, Tennessee
  - University of Texas Southwestern Medical Center at Dallas, Dallas, Texas
  - University of Texas Southwestern Medical Center, Dallas, Texas
- Argentina (2):
  - COIBA Centro de Oncología e Investigación Buenos Aires, Berazategui, Buenos Aires
  - Fundación Investigar, Buenos Aires, Ciudad Autónoma de BuenosAires
- Australia (7):
  - The Tweed Hospital, Tweed Heads, New South Wales
  - Sunshine Coast University Hospital, Birtinya, Queensland
  - Bankstown-Lidcombe Hospital, Bankstown
  - St. George Hospital, Kogarah
  - Box Hill Hospital, Oncology Department, Melbourne
  - Maroondah Hospital, Maroondah Breast Clinic, Melbourne
  - Sydney Adventist Hospital, Wahroonga
- University Hospital Innsbruck - Tyrolean Hospital, Department of Gynecology, Innsbruck, Austria
- Belgium (9):
  - Our Dear Lady Hospital, Aalst Campus, Aalst
  - Institut Jules Bordet - Medical Oncology, Brussels
  - University Hospital Saint-Luc, Brussels
  - Antwerp University Hospital, Edegem
  - Leuven University Hospitals, Leuven
  - Clinic Saint-Joseph, Liège
  - St. Elizabeth Maternity Clinic, Namur
  - AZ Damiaan General Hospital, Sint-Jozef Oncology Center, Ostend
  - Saint-Augustinus Hospital, Wilrijk
- Brazil (13):
  - Centro Regional Integrado de Oncologia, Fortaleza, Ceará
  - Núcleo de Oncologia da Bahia - NOB, Salvador, Estado de Bahia
  - Ensino E Terapia de Inovação Clínica Assistência Multidiciplinar Em Oncologia Ética, Salvador, Estado de Bahia
  - Hospital Araújo Jorge, Associação de Combate ao Câncer em Goiás, Goiânia, Goiás
  - Liga Paranaense de Combate ao Cancer, Hospital Erasto Gaertner, Curitiba, Paraná
  - Instituto de Pesquisas Clinicas para Estudos Multicentricos Hospital Geral de Caxias do Sul, Universidade de Caxias do Sul (IPCEM), Caxias do Sul, Rio Grande do Sul
  - Hospital Sao Lucas da PUCRS, Porto Alegre, Rio Grande do Sul
  - Instituto Joinvillense de Hematologia e Oncologia, Joinville, Santa Catarina
  - Hospital de Cancer de Barretos - Hospital, Barretos, São Paulo
  - Instituto Ribeiraopretano de Combate Ao Cancer - Clinic/Outpatient Facility, Ribeirão Preto, São Paulo
  - Fundação Faculdade Regional de Medicina de São José do Rio Preto, Hospital de Base, São José do Rio Preto, São Paulo
  - Hospital Do Cancer A C Camargo - Hospital, São Paulo
  - Instituto Brasileiro de Controle Do Câncer IBCC, São Paulo
- Canada (13):
  - Tom Baker Cancer Centre, Calgary, Alberta
  - Abbotsford Regional Hospital and Cancer Care Centre, Abbotsford, British Columbia
  - British Columbia Cancer Agency, Kelowna, British Columbia
  - Fraser Health Authority, Surrey, British Columbia
  - Royal Victoria Regional Health Centre, Barrie, Ontario
  - Grand River Hospital, Kitchener, Ontario
  - Ottawa Hospital, Cancer Center, Ottawa, Ontario
  - Toronto East General Hospital, Toronto, Ontario
  - Sunnybrook Health Sciences Center, Odette Cancer Center, Toronto, Ontario
  - St. Michael's Hospital, Toronto, Ontario
  - CHUM Notre Dame Hospital, Montreal, Quebec
  - Montreal General Hospital, Montreal, Quebec
  - Centre hospitalier affilié universitaire de Québec - Hôpital du Saint-Sacrement, Québec, Quebec
- Czechia (3):
  - Masaryk Memorial Cancer Institute, Brno
  - Hospital Novy Jicin, Nový Jičín
  - University Hospital Motol, Comprehensive Oncology Center, Prague
- Sjaelland University Hospital, Næstved, Denmark
- Helsinki University Central Hospital, Department of Oncology, Helsinki, Finland
- France (5):
  - South Lyon Hospital Center, Department of Clinical Hematology and Medical Oncology, Pierre-Bénite, Lyon
  - Center Jean Perrin, Clermont-Ferrand
  - Saint-Louis Hospital, Paris
  - Clinic Sainte Anne, Center for Radiotherapy, Strasbourg
  - Gustave Roussy Oncology Institute, Department of Medicine, Villejuif
- Germany (7):
  - Hematology-Oncology Practice, Augsburg
  - Practice for Oncology Bielefeld, Bielefeld
  - University Hospital Cologne, Breast Center, Clinic of Obstetrics and Gynecology, Cologne
  - University Hospital Schleswig-Holstein, Kiel
  - Otto von Guericke University of Magdeburg, Magdeburg
  - Onkologie Ravensburg, Ravensburg
  - University Hospital Ulm, Ulm
- Hong Kong (6):
  - Prince of Wales Hospital, Shatin, New Territories
  - Queen Elizabeth Hospital, Department of Clinical Oncology, Hong Kong
  - Queen Mary Hospital, Department of Clinical Oncology, Hong Kong
  - Queen Mary Hospital, Department of Oncology, Hong Kong
  - Queen Mary Hospital, Department of Surgery, Hong Kong
  - Tuen Mun Hospital, Hong Kong
- Ireland (2):
  - St. Jame's Hospital, Dublin
  - St. Vincent's University Hospital, Dublin
- Israel (10):
  - Soroka Medical Center, Beersheba
  - Rambam Medical Center, Haifa
  - Shaare Zedek Medical Center, Jerusalem
  - Hadassah Medical Center, Jerusalem
  - Meir Medical Center, Kfar Saba
  - Rabin Medical Center, Belinson Hospital, Petah Tikva
  - Kaplan Medical Center, Department of Oncology, Rehovot
  - Ziv Medical Center, Safed
  - Sourasky Medical Center, Department of Oncology, Tel Aviv
  - Chaim Sheba Medical Center, Tel Litwinsky
- Italy (16):
  - Hospital Papa Giovanni XXIII, Department of Medical Oncology, Bergamo
  - Hospital Cervesi di Cattolica, Department of Oncology, Cattolica
  - University G. D'Annunzio Chieti Pescara, Chieti
  - Scientific Institute of Romagna of the Study and Treatment of Cancer, Meldola
  - IRCCS - Hospital San Raffaele, Department of Medical Oncology, Milan
  - European Institute of Oncology, Milan
  - Azienda Ospedaliero San Gerardo, Monza
  - National Cancer Institute - IRCCS "Fondazione G. Pascale", Naples
  - Hospital Sacro Cuore Don Calabria, Department of Medical Oncology, Negrar
  - Azienda Ospedaliera Regionale San Carlo, Potenza
  - Hospital Bianchi Melacrino Morelli, Reggio Calabria
  - Hospital Infermi Rimini, Unit of Oncology, Rimini
  - University Hospital Campus Bio-Medico, Rome
  - National Cancer Institute Regina Elena, Rome
  - Institute of Cancer Research and Treatment, Torino
  - Hospital Desio and Vimercate, Department of Medical Oncology, Vimercate
- Japan (15):
  - Chiba University Hospital, Chiba, Chiba
  - Kobe City Medical Center General Hospital, Kobe, Hyôgo
  - University of Tsukuba Hospital, Tsukuba, Ibaraki
  - Iwate Medical University Hospital, Morioka, Iwate
  - Tokai University Hospital, Isehara, Kanagawa
  - Kumamoto University Hospital, Kumamoto, Kumamoto
  - Saitama Cancer Centre, Kitaadachi-gun, Saitama
  - JCHO Kurume General Hospital, Fukuoka
  - Gunma University Hospital, Gunma
  - Hiroshima City Hospital, Hiroshima
  - National Hospital Organization Hokkaido Cancer Center, Hokkaido
  - Hakuaikai Medical Corporation Sagara Hospital, Kagoshima
  - Osaka International Cancer Institute, Osaka
  - National Hospital Organization Osaka National Hospital, Ôsaka
  - Toramonon Hospital, Tokyo
- Maastricht University Medical Centre (MUMC), Maastricht, Netherlands
- Portugal (3):
  - Instituto Portugues de Oncologia de Lisboa Francisco Gentil, EPE, Lisbon
  - Centro de Investigação Clinica, Hospital da Luz, Lisbon
  - Instituto Português de Oncologia do Porto Francisco Gentil, E.P.E., Porto
- Russia (3):
  - Federal State Government-Financed Institution: City Clinical Hospital #40, Moscow, Moscow
  - Russian Oncological Research Center n.a. N.N. Blokhin Russian Academy of Medical Sciences, Moscow
  - Tambov Regional Oncological Center, Tambov
- Singapore (7):
  - National University Hospital, Singapore
  - National Cancer Centre Singapore, Department of Medical Oncology, Singapore
  - Raffles Hospital, Singapore
  - Icon Singapore Oncology Consultants Farrer Park Medical Clinic, Singapore
  - Gleneagles Medical Centre, Center for Medical Oncology, Singapore
  - Parkway Cancer Centre, Singapore
  - Johns Hopkins Singapore International Medical Center, Singapore
- South Korea (3):
  - National Cancer Center, Gyeonggi-do
  - Severance Hospital, Seoul
  - Asan Medical Center, Seoul
- Spain (16):
  - Hospital Universitario Vall d'Hebron, Barcelona
  - Consorcio Hospitalario Provincial de Castellon, Castellon
  - Hospital Universitari de Girona Dr. Josep Trueta (ICO Girona), Servicio de Oncologia, Girona
  - Complejo Hospitalario Universitario Insular-Materno Infantil, Las Palmas de Gran Canaria
  - Centro Oncologico MD Anderson, Madrid
  - University Hospital Clinic San Carlos, Servicio de Oncologia Medica, Madrid
  - University Hospital 12 de Octubre, Servicio de Oncologia - Edificio Maternidad, 2ª planta, Madrid
  - Centro Integral Oncologico Clara Campal, Madrid
  - University Hospital Quiron Madrid, Department of Oncology, Madrid
  - Hospital Universitario Virgen de la Arrixaca, Servicio de Oncologia, Murcia
  - Hospital Universitario Son Espases, Palma de Mallorca
  - Hospital Son Llatzer, Servicio de Oncologia, Palma de Mallorca
  - Hospital Universitario Virgen Macarena, Seville
  - University Hospital Virgen del Rocio, Servicio de Oncologia, Seville
  - Hospital Clinico Universitario de Valencia, Servicio de Oncologia, Valencia
  - Hospital Clinico Universitario Lozano Blesa, Servicio de Oncologia, Zaragoza
- Sweden (2):
  - Orebro University Hospital, Department of Oncology, Örebro
  - Uppsala University Hospital, Department of Oncology, Uppsala
- Switzerland (4):
  - Hospital Engeried, Bern
  - University Hospital of Geneva, Geneva
  - Canton Hospital Winterthur, Winterthur
  - Onkozentrum Zurich - Kinik im Park, Zurich
- Taiwan (15):
  - Kaohsiung Chang Gung Memorial Hospital, Kaohsiung City, Province of China
  - Taichung Veterans General Hospital, Breast Center, Taichung, Province of China
  - National Cheng Kung University Hospital, Tainan, Province of China
  - Chi Mei Medical Center - YK Branch, Tainan, Province of China
  - Chi Mei Medical Center - LiouYing Branch, Tainan, Province of China
  - Mackay Memorial Hospital, Taipei, Province of China
  - Tri-Service General Hospital, Taipei, Province of China
  - Changhua Christian Hospital, Changhua, Taiwan, Province of China
  - Buddhist Tzu-Chi General Hospital, Hualien City, Taiwan, Province of China
  - Chung-Ho Memorial Hospital, Kaohsiung City, Taiwan, Province of China
  - Kaohsiung Veterans General Hospital, Kaohsiung City, Taiwan, Province of China
  - Taipei Tzu Chi General Hospital, New Taipei City
  - Kuang Tien General Hospital, Taichung
  - National Taiwan University Hospital, Taipei
  - Taipei Veterans General Hospital, Taipei
- Turkey (Türkiye) (2):
  - Ege University, Bornova, İzmir
  - Marmara University Faculty of Medicine, Istanbul
- United Kingdom (6):
  - Colchester General Hospital, Colchester, Essex
  - Queen Elizabeth Hospital Birmingham, Birmingham, West Midlands
  - Velindre Cancer Centre, Cardiff
  - Calderdale Royal Hospital, Macmillan Unit, Halifax
  - Huddersfield Royal Infirmary, Huddersfield
  - Nottingham City Hospital Campus, Department of Oncology, Nottingham

IPD SHARING:
Plan to Share IPD: Yes
Puma Biotechnology is committed to sharing clinical trial data and information to help physicians and patients make informed treatment decisions, and to help qualified researchers advance scientific knowledge.
  In accordance with legal and regulatory requirements, Puma publishes study protocol information and clinical study results on clinical trial registries, including ClinicalTrials.gov and EU Clinical Trials Register. Puma also publishes information about clinical studies in peer-reviewed scientific journals and shares data in scientific meetings.
  Puma commits to safeguarding confidentiality and patient privacy throughout the clinical trial data and information sharing process. Any patient-level data will be anonymized to protect personally identifiable information.
  Qualified researchers and study participants may submit requests for other study documentation and clinical trial data to clinicaltrials@pumabiotechnology.com for consideration.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Clinical study documents and clinical trial data may be requested by qualified researchers and study participants for studies that have been completed for at least 18 months, and for which the indication of the drug has been approved in the US and/or EU, as applicable. Requests will be accepted for up to 24 months after the criteria described in this section are met.
Access Criteria: Requestors must provide organizational contact information; a detailed research plan, including outcomes; timeline for completion of the research; qualifications of the research team; funding source; and potential conflicts of interest.
  Puma will not provide access to patient-level data if there is a reasonable likelihood that individual patients could be identified, or in cases where confidentiality or consent provisions prohibit transfer of data or information to third parties. Additionally, Puma will not disclose information that jeopardizes intellectual property rights or divulges confidential commercial information.
URL: https://pumabiotechnology.com/data_sharing_policy.html

REFERENCES:
- [Derived] Dai MS, Feng YH, Chen SW, Masuda N, Yau T, Chen ST, Lu YS, Yap YS, Ang PCS, Chu SC, Kwong A, Lee KS, Ow S, Kim SB, Lin J, Chung HC, Ngan R, Kok VC, Rau KM, Sangai T, Ng TY, Tseng LM, Bryce R, Bebchuk J, Chen MC, Hou MF. Analysis of the pan-Asian subgroup of patients in the NALA Trial: a randomized phase III NALA Trial comparing neratinib+capecitabine (N+C) vs lapatinib+capecitabine (L+C) in patients with HER2+metastatic breast cancer (mBC) previously treated with two or more HER2-directed regimens. Breast Cancer Res Treat. 2021 Oct;189(3):665-676. doi: 10.1007/s10549-021-06313-5. Epub 2021 Sep 23. PMID 34553296
- [Derived] Saura C, Oliveira M, Feng YH, Dai MS, Chen SW, Hurvitz SA, Kim SB, Moy B, Delaloge S, Gradishar W, Masuda N, Palacova M, Trudeau ME, Mattson J, Yap YS, Hou MF, De Laurentiis M, Yeh YM, Chang HT, Yau T, Wildiers H, Haley B, Fagnani D, Lu YS, Crown J, Lin J, Takahashi M, Takano T, Yamaguchi M, Fujii T, Yao B, Bebchuk J, Keyvanjah K, Bryce R, Brufsky A; NALA Investigators. Neratinib Plus Capecitabine Versus Lapatinib Plus Capecitabine in HER2-Positive Metastatic Breast Cancer Previously Treated With >/= 2 HER2-Directed Regimens: Phase III NALA Trial. J Clin Oncol. 2020 Sep 20;38(27):3138-3149. doi: 10.1200/JCO.20.00147. Epub 2020 Jul 17. PMID 32678716

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Neratinib Plus Capecitabine | Lapatinib Plus Capecitabine
Started | 307 | 314
Received Treatment | 303 | 311
Completed | 0 | 0
Not Completed | 307 | 314
Not completed — Death | 212 | 240
Not completed — Withdrawal by Subject | 12 | 10
Not completed — Lost to Follow-up | 3 | 0
Not completed — Discontinuation of study by sponsor | 79 | 64
Not completed — Randomized in Error | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Neratinib Plus Capecitabine | Lapatinib Plus Capecitabine | Total
Number analyzed (Participants) | 307 | 314 | 621
Age, Continuous [Mean (Standard Deviation); unit: years] | 55.04 (11.37) | 54.32 (11.36) | 54.67 (11.36)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 307 | 311 | 618
  Male | 0 | 3 | 3
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 40 | 42 | 82
  Not Hispanic or Latino | 256 | 259 | 515
  Unknown or Not Reported | 11 | 13 | 24
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race: Asian | 109 | 105 | 214
  Race: Black or African American | 9 | 15 | 24
  Race: Native Hawaiian or Other Pacific Islander | 1 | 1 | 2
  Race: White | 178 | 177 | 355
  Race: Other | 7 | 10 | 17
  Race: Unknown/Missing | 3 | 6 | 9
Previous HER2 Regimens [Count of Participants; unit: Participants]
  2 | 215 | 215 | 430
  >=3 | 92 | 99 | 191
Disease Location [Count of Participants; unit: Participants]
  Non Visceral | 60 | 61 | 121
  Visceral | 247 | 253 | 500
Hormone Receptor Status [Count of Participants; unit: Participants]
  Negative | 126 | 128 | 254
  Positive | 181 | 186 | 367
Geographic Region [Count of Participants; unit: Participants]
  Europe | 121 | 123 | 244
  North America | 59 | 65 | 124
  Rest of World | 127 | 126 | 253

OUTCOME MEASURES:

1. Primary Outcome: Centrally Assessed Progression Free Survival
Description: Progression Free Survival (PFS), Measured in Months, for Randomized Subjects of the Central Assessment. The time interval from the date of randomization until the first date on which recurrence, progression (per Response Evaluation Criteria in Solid Tumors Criteria (RECIST) v1.1), or death due to any cause, is documented. For subjects without recurrence, progression or death, it is censored at the last valid tumor assessment. Progression is defined using Response Evaluation Criteria in Solid Tumors Criteria (RECIST v1.1), as a 20% increase in the sum of the longest diameter of target lesions, or a measurable increase in a non-target lesion, or the appearance of new lesions. Here, the time to event was reported as the restricted mean survival time. The restricted mean survival time was defined as the area under the curve of the survival function up to 24 months.
Time Frame: From randomization date to recurrence, progression or death, assessed up to 38 months. The result is based on primary analysis data cut.
Population: Randomized ITT Population
Measure: Mean (95% Confidence Interval); unit: months
Arm/Group | Neratinib Plus Capecitabine | Lapatinib Plus Capecitabine
Number analyzed (Participants) | 307 | 314
months | 8.8 [7.8 to 9.8] | 6.6 [5.9 to 7.4]
Statistical Analysis 1: Comparison: Neratinib Plus Capecitabine vs Lapatinib Plus Capecitabine; Test type: Superiority; p = 0.0059, Log Rank; Stratified by hormone receptor status, number of prior HER2-directed regimens in the metastatic setting, and visceral disease vs. non-visceral; Hazard Ratio (HR) = 0.762, 95% CI 2-sided [0.626 to 0.926] — Lapatinib Plus Capecitabine is the reference. Stratified by hormone receptor status, number of prior HER2-directed regimens in the metastatic setting, and visceral disease vs. non-visceral

2. Primary Outcome: Overall Survival
Description: Overall survival (OS) is defined as the time from randomization to death due to any cause, censored at the last date known alive on or prior to the data cutoff employed for the analysis, whichever was earlier. Here, the time to event was reported as the restricted mean survival time. The restricted mean survival time was defined as the area under the curve of the survival function up to 48 months.
Time Frame: From randomization date to death, assessed up to 59 months.The result is based on primary analysis data cut.
Measure: Mean (95% Confidence Interval); unit: months
Arm/Group | Neratinib Plus Capecitabine | Lapatinib Plus Capecitabine
Number analyzed (Participants) | 307 | 314
months | 24.0 [22.1 to 25.9] | 22.2 [20.4 to 24.0]
Statistical Analysis 1: Comparison: Neratinib Plus Capecitabine vs Lapatinib Plus Capecitabine; Test type: Superiority; p = 0.2086, Log Rank; [statistical method as in outcome 1, analysis 1]; Hazard Ratio (HR) = 0.881, 95% CI 2-sided [0.723 to 1.073] — [estimate comment as in outcome 1, analysis 1]

3. Secondary Outcome: Intervention for Symptomatic Metastatic Central Nervous System Disease
Description: Intervention for symptomatic metastatic central nervous system disease is defined as the time from randomization to the first start date of an intervention for symptomatic metastatic CNS disease. Subjects that do not have an intervention for symptomatic metastatic CNS and do not die will be censored at the last date known alive on or prior to the data cutoff. Deaths are treated as competing events. Percentage of participants with intervention for CNS, estimated by cumulative incidence methods. Cumulative incidence methods are the standard way to estimate incidence of an endpoint in the presence of competing risks and censoring.
Time Frame: From randomization date to first intervention for symptomatic metastatic CNS disease, assessed up to 59 months.The result is based on primary analysis data cut.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Neratinib Plus Capecitabine | Lapatinib Plus Capecitabine
Number analyzed (Participants) | 307 | 314
percentage of participants | 22.76 [15.48 to 30.91] | 29.19 [22.54 to 36.14]
Statistical Analysis 1: Comparison: Neratinib Plus Capecitabine vs Lapatinib Plus Capecitabine; Test type: Superiority; p = 0.043, Gray's test; Stratified by hormone receptor status, number of prior HER2-directed regimens in the metastatic setting and visceral disease vs. non-visceral disease

4. Secondary Outcome: Objective Response Rate (ORR) - Central Assessment (ITT Population With Measurable Disease at Screening)
Description: Objective response rate is defined as the percentage of participants demonstrating an objective response during the study. Objective response includes confirmed complete responses (CR) and partial responses (PR) as defined in the RECIST criteria included in the study protocol. The ORR is for Central Assessment for subjects that had measurable disease at screening. Per Response Evaluation Criteria in Solid Tumors Criteria (RECIST v1.0) for target lesions and assessed by MRI: Complete Response (CR), Disappearance of all target lesions; Partial Response (PR), >=30% decrease in the sum of the longest diameter of target lesions; Overall Response (OR) = CR + PR.
Time Frame: From randomization date to first confirmed Complete or Partial Response, whichever came earlier, up to 42 months.The result is based on primary analysis data cut.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Neratinib Plus Capecitabine | Lapatinib Plus Capecitabine
Number analyzed (Participants) | 256 | 270
percentage of participants | 32.8 [27.1 to 38.9] | 26.7 [21.5 to 32.4]
Statistical Analysis 1: Comparison: Neratinib Plus Capecitabine vs Lapatinib Plus Capecitabine; Test type: Superiority; p = 0.1201, Cochran-Mantel-Haenszel; Stratified by hormone receptor status, number of prior HER2-directed regimens in the metastatic setting and visceral disease vs. non-visceral

5. Secondary Outcome: Clinical Benefit Rate (CBR) - Central Assessment (ITT Population With Measurable Disease at Screening)
Description: Clinical benefit rate is the percentage of participants who achieve overall tumor response (confirmed CR or PR) or stable disease (SD) lasting for at least 24 weeks from randomization. The CBR was for Central Assessment for subjects who had Measurable Disease at Screening.
Time Frame: From randomization date to either first confirmed CR or PR or Stable Disease, whichever came earlier, up to 42 months.The result is based on primary analysis data cut.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Neratinib Plus Capecitabine | Lapatinib Plus Capecitabine
Number analyzed (Participants) | 256 | 270
percentage of participants | 44.5 [38.3 to 50.8] | 35.6 [29.8 to 41.6]
Statistical Analysis 1: Comparison: Neratinib Plus Capecitabine vs Lapatinib Plus Capecitabine; Test type: Superiority; p = 0.0328, Cochran-Mantel-Haenszel; [statistical method as in outcome 4, analysis 1]

6. Secondary Outcome: Duration of Response (DOR) - Central Assessment (Population That Had a Response With Measurable Disease at Screening)
Description: The Duration of Response (DOR) is for Central Assessment for the Population that Had a Response with Measurable Disease at Screening.
  Duration of response is measured from the time at which measurement criteria are first met for CR or PR (whichever status is recorded first) until the first date of recurrence or progressive disease (PD) or death is objectively documented, taking as a reference for PD the smallest measurements recorded since enrollment, per RECIST v1.1. This value is censored at the last valid tumor assessment if PD or death has not been documented.
Time Frame: From start date of response after randomization to first PD, up to 33 months.The result is based on primary analysis data cut.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Neratinib Plus Capecitabine | Lapatinib Plus Capecitabine
Number analyzed (Participants) | 84 | 72
months | 8.54 [5.62 to 11.17] | 5.55 [4.21 to 6.41]
Statistical Analysis 1: Comparison: Neratinib Plus Capecitabine vs Lapatinib Plus Capecitabine; Test type: Superiority; p = 0.0004, Log Rank; Hazard Ratio (HR) = 0.495, 95% CI 2-sided [0.332 to 0.736] — Lapatinib Plus Capecitabine is the reference

7. Secondary Outcome: Percentage of Participants With Treatment-Emergent Adverse Events (Adverse Events and Serious Adverse Events)
Description: Adverse Events to be measured are Treatment-Emergent and Serious AEs that occurred on or after first dose of investigational product and up to 28 days after the last dose
Time Frame: From first dose through last dose + 28 days, up to 41 months. The result is based on final data cut.
Population: Safety population: Participants receiving at least 1 dose of investigational product.
Measure: Number; unit: percentage of participants
Arm/Group | Neratinib Plus Capecitabine | Lapatinib Plus Capecitabine
Number analyzed (Participants) | 303 | 311
percentage of participants
  All Treatment-Emergent Adverse Events | 99.7 | 99.4
  Serious Treatment-Emergent Adverse Events | 34.0 | 29.9

ADVERSE EVENTS:
Time Frame: From time of first dose, through 28 days after last dose, assessed up to 41 months.
Description: Safety population: Participants receiving at least 1 dose of investigational product.
  All-Cause Mortality was monitored/assessed for all randomized participants. Serious and Other Adverse Events were monitored/assessed only in the safety population
  For All-Cause Mortality and Serious/Other Adverse Events, the result is based on final data cut.
Arm/Group | Neratinib Plus Capecitabine | Lapatinib Plus Capecitabine
All-Cause Mortality (participants affected / at risk) | 219/307 | 243/314
Serious Adverse Events (participants affected / at risk) | 103/303 | 93/311
Other Adverse Events (participants affected / at risk) | 301/303 | 309/311
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Neratinib Plus Capecitabine (N=303) | Lapatinib Plus Capecitabine (N=311)
Anaemia (Blood and lymphatic system disorders) | 1 | 2
Febrile neutropenia (Blood and lymphatic system disorders) | 1 | 3
Neutropenia (Blood and lymphatic system disorders) | 1 | 0
Acute myocardial infarction (Cardiac disorders) | 0 | 1
Atrial fibrillation (Cardiac disorders) | 1 | 0
Cardiac arrest (Cardiac disorders) | 0 | 1
Cardiac tamponade (Cardiac disorders) | 1 | 1
Cardiomyopathy (Cardiac disorders) | 1 | 0
Palpitations (Cardiac disorders) | 2 | 0
Pericardial effusion (Cardiac disorders) | 1 | 1
Tachycardia (Cardiac disorders) | 0 | 1
Vertigo (Ear and labyrinth disorders) | 1 | 0
Chorioretinopathy (Eye disorders) | 1 | 0
Abdominal distension (Gastrointestinal disorders) | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 1 | 5
Abdominal pain upper (Gastrointestinal disorders) | 2 | 0
Ascites (Gastrointestinal disorders) | 0 | 2
Constipation (Gastrointestinal disorders) | 3 | 1
Diarrhoea (Gastrointestinal disorders) | 22 | 13
Gastric ulcer (Gastrointestinal disorders) | 2 | 1
Gastritis (Gastrointestinal disorders) | 0 | 1
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 | 0
Nausea (Gastrointestinal disorders) | 7 | 6
Pancreatitis (Gastrointestinal disorders) | 2 | 0
Pancreatitis acute (Gastrointestinal disorders) | 1 | 0
Stomatitis (Gastrointestinal disorders) | 1 | 1
Varices oesophageal (Gastrointestinal disorders) | 1 | 0
Vomiting (Gastrointestinal disorders) | 9 | 6
Abasia (General disorders) | 0 | 1
Asthenia (General disorders) | 1 | 2
Chest pain (General disorders) | 1 | 0
Fatigue (General disorders) | 2 | 0
General physical health deterioration (General disorders) | 1 | 2
Malaise (General disorders) | 0 | 1
Multiple organ dysfunction syndrome (General disorders) | 1 | 0
Non-cardiac chest pain (General disorders) | 1 | 2
Oedema (General disorders) | 1 | 0
Pyrexia (General disorders) | 3 | 0
Suprapubic pain (General disorders) | 0 | 1
Bile duct obstruction (Hepatobiliary disorders) | 1 | 0
Hepatic failure (Hepatobiliary disorders) | 1 | 1
Hepatic mass (Hepatobiliary disorders) | 1 | 0
Hepatitis fulminant (Hepatobiliary disorders) | 0 | 1
Jaundice (Hepatobiliary disorders) | 0 | 2
Jaundice cholestatic (Hepatobiliary disorders) | 1 | 1
Hypersensitivity (Immune system disorders) | 1 | 0
Abdominal infection (Infections and infestations) | 1 | 0
Atypical pneumonia (Infections and infestations) | 1 | 0
Bacteraemia (Infections and infestations) | 1 | 1
Catheter site infection (Infections and infestations) | 0 | 1
Cellulitis (Infections and infestations) | 4 | 5
Enterocolitis infectious (Infections and infestations) | 0 | 1
Epiglottitis (Infections and infestations) | 1 | 0
Erysipelas (Infections and infestations) | 0 | 1
Gastroenteritis (Infections and infestations) | 1 | 0
Influenza (Infections and infestations) | 0 | 2
Lung infection (Infections and infestations) | 2 | 0
Paronychia (Infections and infestations) | 1 | 0
Pneumonia (Infections and infestations) | 6 | 5
Pneumonia bacterial (Infections and infestations) | 1 | 0
Respiratory tract infection (Infections and infestations) | 1 | 1
Sepsis (Infections and infestations) | 1 | 4
Septic shock (Infections and infestations) | 0 | 1
Soft tissue infection (Infections and infestations) | 0 | 1
Streptococcal sepsis (Infections and infestations) | 1 | 0
Tooth infection (Infections and infestations) | 0 | 1
Upper respiratory tract infection (Infections and infestations) | 2 | 0
Urinary tract infection (Infections and infestations) | 3 | 1
Urosepsis (Infections and infestations) | 0 | 1
Viral upper respiratory tract infection (Infections and infestations) | 0 | 1
Wound infection (Infections and infestations) | 0 | 1
Fall (Injury, poisoning and procedural complications) | 2 | 2
Femur fracture (Injury, poisoning and procedural complications) | 1 | 1
Fracture (Injury, poisoning and procedural complications) | 0 | 1
Head injury (Injury, poisoning and procedural complications) | 1 | 0
Hip fracture (Injury, poisoning and procedural complications) | 1 | 0
Humerus fracture (Injury, poisoning and procedural complications) | 2 | 0
Seroma (Injury, poisoning and procedural complications) | 1 | 0
Blood bilirubin increased (Investigations) | 0 | 3
Blood potassium increased (Investigations) | 0 | 1
Liver function test increased (Investigations) | 0 | 1
Weight decreased (Investigations) | 2 | 0
Decreased appetite (Metabolism and nutrition disorders) | 1 | 0
Dehydration (Metabolism and nutrition disorders) | 4 | 5
Hypercalcaemia (Metabolism and nutrition disorders) | 1 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 2 | 4
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 1
Hypophosphataemia (Metabolism and nutrition disorders) | 0 | 2
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 2
Bone pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 | 1
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Osteonecrosis of jaw (Musculoskeletal and connective tissue disorders) | 0 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 4
Pathological fracture (Musculoskeletal and connective tissue disorders) | 0 | 1
Brain neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Endometrial cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Intracranial tumour haemorrhage (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Malignant pleural effusion (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Metastases to bone (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Metastases to central nervous system (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 6 | 2
Papillary thyroid cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Pericarditis malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Tumour compression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Tumour haemorrhage (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 2
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Amnesia (Nervous system disorders) | 0 | 1
Aphasia (Nervous system disorders) | 0 | 2
Ataxia (Nervous system disorders) | 0 | 1
Brain oedema (Nervous system disorders) | 0 | 2
Cerebellar syndrome (Nervous system disorders) | 1 | 0
Cerebral haematoma (Nervous system disorders) | 1 | 0
Cerebral infarction (Nervous system disorders) | 0 | 1
Cerebrovascular accident (Nervous system disorders) | 1 | 0
Dizziness (Nervous system disorders) | 1 | 2
Haemorrhage intracranial (Nervous system disorders) | 0 | 1
Headache (Nervous system disorders) | 1 | 6
Hemiparesis (Nervous system disorders) | 1 | 1
Hypoaesthesia (Nervous system disorders) | 0 | 1
Intracranial pressure increased (Nervous system disorders) | 2 | 0
Lethargy (Nervous system disorders) | 1 | 1
Nerve root compression (Nervous system disorders) | 1 | 0
Neurological decompensation (Nervous system disorders) | 0 | 1
Neuropathy peripheral (Nervous system disorders) | 1 | 0
Paraparesis (Nervous system disorders) | 1 | 0
Presyncope (Nervous system disorders) | 1 | 0
Seizure (Nervous system disorders) | 4 | 3
Spinal cord oedema (Nervous system disorders) | 1 | 0
Subarachnoid haemorrhage (Nervous system disorders) | 0 | 1
Syncope (Nervous system disorders) | 1 | 0
Tonic convulsion (Nervous system disorders) | 0 | 1
Confusional state (Psychiatric disorders) | 1 | 1
Delirium (Psychiatric disorders) | 0 | 1
Disorientation (Psychiatric disorders) | 1 | 0
Mental status changes (Psychiatric disorders) | 0 | 1
Acute kidney injury (Renal and urinary disorders) | 7 | 1
Hydronephrosis (Renal and urinary disorders) | 0 | 1
Renal failure (Renal and urinary disorders) | 1 | 0
Vaginal haemorrhage (Reproductive system and breast disorders) | 1 | 0
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 | 3
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 10 | 11
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 2 | 7
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 1 | 1
Skin necrosis (Skin and subcutaneous tissue disorders) | 0 | 1
Hypotension (Vascular disorders) | 0 | 2
Shock (Vascular disorders) | 0 | 1
Vena cava thrombosis (Vascular disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Neratinib Plus Capecitabine (N=303) | Lapatinib Plus Capecitabine (N=311)
Anaemia (Blood and lymphatic system disorders) | 45 | 50
Neutropenia (Blood and lymphatic system disorders) | 23 | 16
Abdominal distension (Gastrointestinal disorders) | 25 | 9
Abdominal pain (Gastrointestinal disorders) | 37 | 42
Abdominal pain upper (Gastrointestinal disorders) | 18 | 28
Constipation (Gastrointestinal disorders) | 95 | 40
Diarrhoea (Gastrointestinal disorders) | 248 | 205
Dry mouth (Gastrointestinal disorders) | 15 | 18
Dyspepsia (Gastrointestinal disorders) | 20 | 29
Nausea (Gastrointestinal disorders) | 161 | 130
Stomatitis (Gastrointestinal disorders) | 63 | 83
Vomiting (Gastrointestinal disorders) | 138 | 95
Asthenia (General disorders) | 36 | 34
Fatigue (General disorders) | 102 | 97
Oedema peripheral (General disorders) | 16 | 21
Pyrexia (General disorders) | 32 | 32
Paronychia (Infections and infestations) | 35 | 49
Upper respiratory tract infection (Infections and infestations) | 26 | 14
Urinary tract infection (Infections and infestations) | 27 | 12
Viral upper respiratory tract infection (Infections and infestations) | 20 | 23
Alanine aminotransferase increased (Investigations) | 27 | 22
Aspartate aminotransferase increased (Investigations) | 29 | 28
Blood bilirubin increased (Investigations) | 18 | 34
Weight decreased (Investigations) | 60 | 41
Decreased appetite (Metabolism and nutrition disorders) | 107 | 67
Dehydration (Metabolism and nutrition disorders) | 14 | 16
Hypokalaemia (Metabolism and nutrition disorders) | 35 | 41
Arthralgia (Musculoskeletal and connective tissue disorders) | 29 | 20
Back pain (Musculoskeletal and connective tissue disorders) | 30 | 22
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 19 | 14
Pain in extremity (Musculoskeletal and connective tissue disorders) | 25 | 21
Dizziness (Nervous system disorders) | 43 | 30
Dysgeusia (Nervous system disorders) | 17 | 13
Headache (Nervous system disorders) | 32 | 50
Insomnia (Psychiatric disorders) | 20 | 23
Cough (Respiratory, thoracic and mediastinal disorders) | 41 | 34
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 19 | 26
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 13 | 20
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 13 | 23
Dry skin (Skin and subcutaneous tissue disorders) | 20 | 15
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 139 | 175
Pruritus (Skin and subcutaneous tissue disorders) | 26 | 25
Rash (Skin and subcutaneous tissue disorders) | 31 | 69
Skin fissures (Skin and subcutaneous tissue disorders) | 9 | 19
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 7 | 17

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2014-02-13): https://cdn.clinicaltrials.gov/large-docs/73/NCT01808573/Prot_000.pdf
  • Statistical Analysis Plan (2018-11-14): https://cdn.clinicaltrials.gov/large-docs/73/NCT01808573/SAP_001.pdf